CLINICAL TRIAL: NCT00504010
Title: The Role of Arnica on Muscle Pain Following Eccentric Exercise
Acronym: Arnica
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: David W. Bauer, MD, Memorial Hermann Healthcare System
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: HSC-MH-07-0202
Record Dates: First submitted 2007-07-17; First posted 2007-07-19 (Estimated); Last update posted 2009-01-07 (Estimated); Status verified 2009-01

CONDITIONS: Muscles; Exercise; Arnica
Keywords: arnica; muscle soreness; exercise; eccentric
MeSH Terms: conditions — Motor Activity; Myalgia | interventions — Arnicae flos extract

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): arnica containing cream
  Interventions: Drug: Arnica Montana
- 2 (Placebo Comparator): carrier cream without arnica
  Interventions: Drug: placebo cream

INTERVENTIONS:
Drug: Arnica Montana — Applied to lower extremity once a day for 3 days
  Arms: 1
Drug: placebo cream — placebo cream applied to leg daily for 3 days
  Arms: 2

SUMMARY:
Arnica in a topical gel formulation will be compared to a placebo to determine whether it decreases muscle soreness following leg exercise when applied to the legs.

DETAILED DESCRIPTION:
Design: The design is a randomized, placebo-controlled, double-blind trial. Each participant will receive 2 containers of gel. One container will be marked "LEFT" and one "RIGHT." One container will contain a commercially available arnica gel formulation, and the other will contain a placebo gel, identical in appearance to the arnica. Subjects will not know which container contains which product. Each participant will also be given a form containing an analog pain scale for each leg. The participant will rate his or her pain in each leg separately on the day before exercise. Each subject will then be asked to perform calf raises using the following protocol:

* The participant removes shoes.
* Active range of motion of the ankle is measured bilaterally using a goniometer.
* He or she places the metatarsal portion of his or her foot on a step that is 7 inches above the floor. Handrails are provided for safety and comfort
* He or she then performs heel lifts by rising up on the stair using the foot on the stair, holds this for 2 seconds, then maximally dorsiflexes the foot for a count of 2 seconds. A metronome set to generate a tone every 2 seconds guides the pace of this.
* This is repeated 25 times, or until the subject is unable to complete a full cycle.
* He or she then performs the same sequence using the other leg.
* A second set of 20 repetitions is performed in each leg, followed by a final 15 repetitions.
* The gel is applied immediately after exercise to both lower legs. Subjects are instructed not to wash off the leg for at least one hour after application.
* The pain score is completed for each leg 24 hours later, and the gel is applied to each leg. Again, subjects are instructed to leave the gel undisturbed for at least one hour.
* Approximately 48 hours later the subject returns for measurement of ankle range of motion, again completes a pain score and applies the gel for a final time. Subjects are instructed to leave the gel on the legs for at least one hour.
* To measure muscle tenderness, a 1cm sphere is placed on the subject's mid-calf, and compressed by a standardized 5 pound weight. The subject provides a tenderness score for each leg using the same pain score.
* A final pain score is completed by each subject at approximately 72 hours.

Neither subjects nor the researchers doing the data collection or analysis will know which gel is associated with which formulation (placebo vs. Arnica). Controls are within-subjects.

ELIGIBILITY:
Inclusion Criteria:

* age 18 or older
* two fully functional legs

Exclusion Criteria:

* allergy or sensitivity to the ester family
* open wound or inflammatory condition on legs
* chronic or acute leg pain
* neuropathy involving one or both legs

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2007-08; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Muscle soreness | 24 - 72 hours

SECONDARY OUTCOMES:
Muscle tenderness | 48 hours
Range of motion of ankle joint | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: David W Bauer, MD, Principal Investigator — Memorial Hermann
Locations (1):
- Memorial Family Medicine, Houston, Texas, United States